CLINICAL TRIAL: NCT00440596
Title: Mindfulness Based Stress Reduction for High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Joel Hughes, Professor, Kent State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT002698-01A2 (NIH)
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Mindfulness-Based Stress Reduction; Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness based stress reduction (Experimental): Mindfulness based stress reduction
  Interventions: Behavioral: Mindfulness based stress reduction
- Progressive Muscle Relaxation (Active Comparator): Progressive Muscle Relaxation
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction — 8 weeks group MBSR
  Arms: Mindfulness based stress reduction
Behavioral: Progressive Muscle Relaxation — 8 weeks PMR in group format
  Arms: Progressive Muscle Relaxation

SUMMARY:
Nearly 60 million adults in the United States have high blood pressure (BP) in the pre-hypertension (SBP 120-139 or DBP 80-89). Hypertension is estimated to account for 1 in 8 deaths in the world, and in the US the direct and indirect costs of high BP are estimated to reach $59.7 billion in 2005. JNC-7 guidelines recommend lifestyle modifications for prehypertension, followed by antihypertensive medication if BP progresses to Stage I hypertension. Mindfulness-based Stress Reduction (MBSR) is an increasingly popular practice that has been purported to alleviate stress and treat certain health conditions. Some stress management therapies and one meditation therapy (e.g., Transcendental Meditation) have shown promise in reducing elevated BP, but MBSR has not been evaluated as a treatment for high BP. When added to lifestyle modification advice, MBSR may be an appropriate complementary treatment for prehypertension. However, prior to a large randomized clinical trial of MBSR for prehypertension and/or hypertension, pilot data is necessary to provide preliminary evidence of a treatment effect and to evaluate feasibility. This feasibility randomized clinical trial of MBSR for unmedicated prehypertension will provide preliminary evidence to support a larger randomized clinical trial by evaluating the feasibility and safety of MBSR as a complementary treatment for high BP and by documenting any treatment effect. Sixty patients with unmedicated BP in the range of SBP 120-139 mm Hg or DBP 80-89 mm Hg will be randomly assigned to MBSR or a progressive muscle relaxation control condition. All patients will receive lifestyle modification advice. Patients will complete 8 weeks of MBSR delivered in a group format by an experienced psychologist trained in MBSR or 8 weeks of progressive muscle relaxation training matched for therapist contact and homework. Patients BP will be assessed prior to randomization and following treatment by researchers blind to treatment assignment. Accrual rates, acceptance of randomization, treatment adherence, treatment fidelity, and patient satisfaction with treatment will be evaluated.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* prehypertension
* 30-60 years of age

Exclusion Criteria:

* normal BP
* hypertension
* pregnancy
* smoking
* use of antihypertensive medication

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2006-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel W Hughes, Ph.D., Principal Investigator — Kent State University
Locations (1):
- Summa Health System, Akron, Ohio, United States

REFERENCES:
- [Derived] Hughes JW, Fresco DM, Myerscough R, van Dulmen MH, Carlson LE, Josephson R. Randomized controlled trial of mindfulness-based stress reduction for prehypertension. Psychosom Med. 2013 Oct;75(8):721-8. doi: 10.1097/PSY.0b013e3182a3e4e5. PMID 24127622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 248 Assessed for eligibility 192 excluded
Pre-assignment Details: 181 did not meet inclusion criteria 11 did not consent to participate
Groups:
- MBSR: Mindfulness based stress reduction
- Progressive Muscle Relaxation: Progressive Muscle Relaxation 8 weeks group treatment
Period: Overall Study
Arm/Group | MBSR | Progressive Muscle Relaxation
Started | 28 | 28
Completed | 21 | 17
Not Completed | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBSR | Progressive Muscle Relaxation | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 56
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (5.8) | 49.5 (7.2) | 50.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: SBP
Time Frame: 12 weeks
Population: 56 participatns intent to treat
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | MBSR | Progressive Muscle Relaxation
Number analyzed (Participants) | 28 | 28
mm Hg | 130.2 (6.3) | 128.8 (6.3)

2. Primary Outcome: DBP
Description: Clinic BP
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | MBSR | Progressive Muscle Relaxation
Number analyzed (Participants) | 28 | 28
mm Hg | 77.3 (4.8) | 78.3 (6.1)

ADVERSE EVENTS:
Arm/Group | MBSR | Progressive Muscle Relaxation
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No